CLINICAL TRIAL: NCT06639139
Title: The Effectiveness of Cognitive-Functional Remote Group Intervention (Cog-Fun RG) for Adults with Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Adina Maeir, Prof. Adina Maeir, School of Occupational Therapy, Hebrew University, Hebrew University of Jerusalem
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 10032020
Record Dates: First submitted 2024-10-06; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: ADHD
Keywords: Occupational Therapy; Executive Functions; Remote Group Therapy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CogFun RG occupational therapy (Experimental): Occupational Therapy Remote Group Intervention . 21 weekly, online group sessions (4-6 participants in each group), lasting 90 minutes. Sessions are structured, comprising opening, collaborative learning, and summary. Session topics include learning about ADHD as a biological disorder of executive functioning, understanding the impact of ADHD on daily life, discovering strategies for coping with ADHD through exploration of life experiences, and preparing for future self-management.
  Interventions: Behavioral: CogFun RG occupational therapy
- Waitlist Control Group (No Intervention): Waiting list, no intervention. After waitlist period will receive the same intervention as the first arm

INTERVENTIONS:
Behavioral: CogFun RG occupational therapy — 21 weekly, online group sessions (4-6 participants in each group), lasting 90 minutes. Sessions are structured, comprising opening, collaborative learning, and summary. Session topics include learning about ADHD as a biological disorder of executive functioning, understanding the impact of ADHD on daily life, discovering strategies for coping with ADHD through exploration of life experiences, and preparing for future self management
  Arms: CogFun RG occupational therapy

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of Cognitive-Functional Remote Group intervention (Cog-Fun RG).

The main questions of this study are 1. will participants demonstrate improvements in their executive functioning and quality of life after receiving the intervention, compared to waitlist controls. In addition, the investigators will examine if the waitlist group will demonstrate similar gains in these outcomes after receiving the same intervention.

the investigators will compare between the intervention group to the waiting list group to examine the effect of the intervention.

The participants will be allocated into two groups: an intervention group and a waiting list group.

The intervention group will receive the the Cog-Fun RG intervention, which includes 21 weekly group sessions, each lasting 90 minutes. the participants will be required to complete questionnaires at several time points: pre-post the intervention, as well as three months, six months, and one year after the intervention.

The waiting list controls will be required to complete questionnaires at several time points: pre-post waiting period, and then after the intervention, as well as three months, six months, and one year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self Reported ADHD diagnoses

Exclusion Criteria:

* Self Reported other major health condition that impedes daily functioning

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The adult ADHD quality of life scale | at baseline, immediately after the intervention, immediately after the waiting period and 3 months after the intervention follow up
  Questionnaire with 29 questions relating to productivity, life outlook, relationships and psychological health. each question is rated on a 5 point scale. Raw scores are transformed to a 1-100 scale. higher scores indicate higher quality of life. The assessment will be conducted at baseline, immediately after the intervention, immediately after the waiting period and 3 months after the intervention follow up.

SECONDARY OUTCOMES:
Behavioral Rating Inventory of Executive Functions (BRIEF) Adult Self -Report | at baseline, immediately after the intervention, immediately after the waiting period.
  Self-report questionnaire for adults evaluates Executive Functions (EF) in everyday contexts. Comprising 75 items rated on a three-point scale (1 = never, 2 = occasionally, 3 = often), the questionnaire categorizes items into nine scales representing distinct EF domains, along with two primary indices. The first, the Behavioral Regulation Index (BRI), encompasses inhibition, shifting, emotional regulation, and behavioral monitoring. The second, the Metacognitive Index (MI), includes working memory, initiation, planning/organization, task monitoring, and organization of materials. These indices contribute to a composite summary score known as the Global Executive Composite (GEC). raw scores are transposed to T-scores based on norms. The assessment will be conducted pre-post the intervention. Higher scores indicating greater difficulty with EF; a score of 65 or above signifies clinical impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebrew University, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No
currently we do not have such a plan we will be happy to consider this in the future

REFERENCES:
- [Background] Galili-Simhon S, Maeir A. Cognitive Functional Remote Group intervention for adults with attention deficit hyperactivity disorder: A feasibility study. Br J Occup Ther. 2023 Oct;86(10):686-696. doi: 10.1177/03080226231177842. Epub 2023 Jun 5. PMID 40337196
- [Background] Kastner L, Velder-Shukrun Y, Bonne O, Bar-Ilan RT, Maeir A. Pilot Study of the Cognitive-Functional Intervention for Adults (Cog-Fun A): A Metacognitive-Functional Tool for Adults With Attention Deficit Hyperactivity Disorder. Am J Occup Ther. 2022 Mar 1;76(2):7602205070. doi: 10.5014/ajot.2022.046417. PMID 35258515